CLINICAL TRIAL: NCT01525472
Title: Accelerated Aging of the Cells of Visceral Adipose Tissue in Morbid Obese Subjects: Involvement in Diseases Associated With Obesity (Viellissement accéléré Des Cellules du Tissu Adipeux viscéral Chez Les obèses Morbides: Implication Dans Les Pathologies associées à l'obésité)
Brief Title: Accelerated Aging of the Cells of Visceral Adipose Tissue in Morbid Obese Subjects
Acronym: SENAPID
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C11-18'; 2011-A01070-41 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Morbid Obesity
Keywords: obesity; adipose tissue; angiogenesis; senecence
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — adipose tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Numerous epidemiological studies clearly showed the relationship between the excessive growth of visceral adipose tissue and risk of developing insulin resistance, type 2 diabetes and other cardiovascular risk factors. However, the mechanisms contributing to the deleterious role of visceral adipose tissue remain to be elucidated. Several observations suggest that adipose tissue depots exhibit distinct metabolic and secretory capacities according to their locations. We have recently shown that visceral fat depots display higher immuno-inflammatory cells infiltration than that of subcutaneous fat. In addition, the endothelial cells of visceral compared to subcutaneous adipose tissues express a pro-inflammatory phenotype and several markers related to aging. Finally, we have shown that visceral adipocyte-derived secretions promote the endothelial cell senescence in an extent higher than subcutaneous adipocyte-derived products. These data suggest that senescence 1) might be a phenomenon related to the location and therefore the microenvironment of adipose tissue and 2) might be responsible for an abnormal activation of proinflammatory response, favouring the development of metabolic and secretory dysfunction of adipose tissue in obesity. Our working hypothesis, based on these observations, is that the visceral adipose tissue provides a microenvironment that promotes accelerated aging. This senescence may be responsible for the establishment of an inflammatory reaction, alteration of the metabolic activity and adipocyte differentiation capacity of progenitor cells leading to the development of obesity associated diseases.

The proposed project is a descriptive cross-sectional pathophysiological study .The aims are 1) to better define the process of senescence in human adipose tissue, 2) to precise the mechanisms and 3) to analyse the cellular and functional consequences of aging on inflammation, adipose tissue development and metabolism. 200 morbidly obese candidates for bariatric surgery will be studied. The collection of clinical and laboratory data and the collection of biological samples (plasma, blood cells and subcutaneous and visceral adipose tissues) will be made at the inclusion and during surgery (obesity center, Hôpital Louis Mourier). Analyses of adipose tissue will be performed at INSERM U1048 and will focus on in vitro approaches of the cells of the adipose tissues (mature adipocytes, endothelial cells, progenitor cells and immuno-inflammatory cells).

This project will permit to better understand the pathogenicity associated with the excessive growth of visceral adipose tissue and may reveal new therapeutic targets to limit obesity-associated pathologies.

DETAILED DESCRIPTION:
Main objective: The main objectives are 1) to compare the state of senescence of subcutaneous versus visceral adipose tissues and 2) to define the senescent cell populations in subcutaneous and visceral adipose tissues in morbidly obese patients.

Secondary objectives: Secondary objectives are 1) to precise whether the state of senescence is attributable to microenvironment, 2) to determine the impact of aging on cellular function, 3) to establish a link between the state of senescence of subcutaneous and visceral adipose tissues and obesity-associated pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 y
* Social security insurance
* Candidate for bariatric surgery based on criteria established by international experts (BMI> 40 or> 35 kg / m² with comorbidities, after failure of multidisciplinary care for a period of at least 1 year)
* Patient having signed an informed consent

Exclusion criteria

* Subject under guardian ship, curator ship or judicial protection.
* Subject taking anti-inflammatory and / or non-steroidal drug
* Current immunosuppressive therapy or interrupted for less than six months
* malignancy or severe inflammatory disease evolving
* Positive HIV serology and / or HBV and / or HCV
* Current pregnancy
* medical or psychiatric contraindication for bariatric surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospital center
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2012-02-13 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Louis Mourier, Colombes, France